CLINICAL TRIAL: NCT06012669
Title: A Randomized, Double-blind, Controlled, Parallel-arm Trial to Assess the Effects of Lactoferrin at Two Doses vs. Active Control on Markers of Immune Function in Healthy Adults
Brief Title: Effects of Lactoferrin at Two Doses vs. Active Control on Markers of Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Helaina Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2305
Record Dates: First submitted 2023-08-16; First posted 2023-08-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Immune Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose (Experimental): 0.34 g Recombinant Human Lactoferrin
  Interventions: Dietary Supplement: Low dose Human Lactoferrin
- High Dose (Experimental): 3.4 g Recombinant Human Lactoferrin
  Interventions: Dietary Supplement: High dose Human Lactoferrin
- Active Control (Active Comparator): 3.4 g Bovine Lactoferrin
  Interventions: Dietary Supplement: Active Control Bovine Lactoferrin

INTERVENTIONS:
Dietary Supplement: High dose Human Lactoferrin — Dietary Supplement and Food Ingredient
  Arms: High Dose
Dietary Supplement: Low dose Human Lactoferrin — Dietary Supplement and Food Ingredient
  Arms: Low Dose
Dietary Supplement: Active Control Bovine Lactoferrin — Dietary Supplement and Food Ingredient
  Arms: Active Control

SUMMARY:
The purpose of this study is to evaluate the impact of 28-day supplementation with high-dose human recombinant lactoferrin, low-dose human recombinant lactoferrin, and an active control product formulated with bovine lactoferrin on indicators of immunity in healthy males and females.

DETAILED DESCRIPTION:
Samples will be retained for possible analyses such as lactoferrin absorption, distribution, metabolism, and excretion (ADME) and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is male or premenopausal female (approximately half males and half females), 18 to 45 years of age, inclusive.
2. Individual has a BMI of ≥18.50 and <30.00 kg/m2.
3. Individual is judged to be in good health based on medical history and routine laboratory tests.
4. Individual agrees to abstain from alcohol consumption and vigorous physical activity for at least 24 h prior to all test visits. According to the World Health Organization (WHO), vigorous physical activity may include running, fast cycling, fast swimming, or moving heavy objects.
5. Individual understands the study procedures, and is willing to complete them, and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Individual is unwilling to avoid consumption of all dietary supplements (other than provided study products and multivitamin/mineral/calcium supplements) within 14 days of visit (day 0) and throughout the study period.
2. Individual is a chronic user of nicotine products.
3. Individual has a score <7 on the Vein Access Scale.
4. Individual has a positive test for illicit drugs on the urine drug screen.
5. Individual has a clinically significant medical condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
6. Individual has an autoimmune disorder (e.g., type 1 diabetes, rheumatoid arthritis, Graves disease, multiple sclerosis, lupus, etc.).
7. Individual has a gastrointestinal condition that would potentially interfere with absorption of the study product (e.g., inflammatory bowel disease, celiac disease, history of gastric bypass surgery, chronic gastritis).
8. Individual has used medication or over-the-counter products (including herbal and dietary supplements) that, in the opinion of the investigator, could interfere with the absorption and metabolism of lactoferrin or affect inflammatory or immune function markers including, but not limited to, aspirin, anti-inflammatories, antacids, histamine 2 receptor antagonists, laxatives, stool softeners, and proton-pump inhibitors.
9. Individual has had a weight change of ±4.5 kg (10 lbs.) in the previous 3 months.
10. Individual has extreme dietary habits (e.g., Atkins, vegan, very low carbohydrate diet).
11. Individual has history of bariatric surgery, is currently taking a weight loss drug, or is actively attempting to lose or gain body weight.
12. Individual has an active infection or signs/symptoms of an infection. Test visits will be rescheduled to allow the subject to be symptom-free of any type of systemic infection for at least five days.
13. Individual has recent use of antibiotics (within 7 days of visit 2, day 0) and throughout the study period. The test days will be rescheduled to allow the subject to wash out the antibiotic for at least 7 days.
14. Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg) at screening.
15. Individual has a history of cancer in the prior 2 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
16. Individual has an allergy or sensitivity to any components of the study products.
17. Individual has an allergy or sensitivity to yeast.
18. Individual is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
19. Individual has been exposed to any non-registered drug product within 30 days of the screening visit.
20. Individual has a current or recent history (past 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
21. Individual has a condition the Investigator believes would interfere with his/her/their ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Antibodies | 0, 8 weeks
  Change from baseline in anti-lactoferrin antibodies

SECONDARY OUTCOMES:
Markers of Immune Function | 0, 4 weeks, 8 weeks, 12 weeks
  Change from baseline in markers of Immune Function (such as biomarkers of inflammation)
Markers of Immune Function | 0, 8 weeks
  Change from baseline in markers of Immune Function (such as T-cell responses to lactoferrin and related peptides)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research & Consulting, LLC
Locations (2):
- United States (2):
  - Suncoast Research, Miami, Florida
  - Health Awareness, Port Saint Lucie, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson RD, Guarneiri LL, Adams CG, Wilcox ML, Clark AJ, Rudemiller NP, Maki KC, Malinczak CA. A Randomized, Double-Blind, Controlled Trial to Assess the Effects of Lactoferrin at Two Doses vs. Active Control on Immunological and Safety Parameters in Healthy Adults. Int J Toxicol. 2025 Jan-Feb;44(1):12-28. doi: 10.1177/10915818241293723. Epub 2024 Oct 28. PMID 39465888